CLINICAL TRIAL: NCT07209709
Title: Comparison of the Effects of Dual Task Training and Action Observation Therapy Given to Geriatric Individuals
Brief Title: Should Dual Task Training or Action Observation Therapy be Used in Geriatric Individuals?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Gizem Gul Turan, Phd Student and Lecturer, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Geriatric Individuals
Record Dates: First submitted 2025-09-22; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Comparison of the Effects of Different Therapies in Geriatric Individuals
Keywords: Action Observation Therapy; Physical Activity; Geriatric Individuals; Dual Task Training; Rehabilitation
MeSH Terms: conditions — Motor Activity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Dual Task Training (DTT) Group: Individuals in this group will participate in exercise sessions consisting of cognitive tasks combined with conventional exercises, 3 days a week, for a total of 8 weeks, under the supervision of a physical therapist.
  Action Observation Therapy (EGT) Group: Individuals in this group will watch exercises on a computer screen in 3 periods (in bed, sitting, and standing) 3 days a week, for a total of 8 weeks. Each exercise in each period will be monitored for 2 minutes, and each exercise session will be performed under the supervision of a physiotherapist for 1 minute. There will be a 1-minute break between each period.
  Control Group (CG): Individuals in this group will participate in conventional exercise sessions 3 days a week, for a total of 8 weeks, under the supervision of a physiotherapist.
  Each session will last an average of 40-50 minutes.
Masking Description: This is an open-label randomized controlled trial. Due to the nature of the exercise interventions, no masking was performed for participants, care providers, investigators, or outcome assessors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dual Task Training (DTT) Group (Experimental): Cognitive functions will be assessed with the "Mini Mental State Test" and "Clock Drawing Test", balance and walking with the "Tinetti Balance and Walking Test", functional mobility with the "Timed Up and Go Test", muscle strength with a handheld dynanometer and "5-times chair sit-to-stand test", flexibility with the "sit-and-reach flexibility test", quality of life with the "CASP-19 Scale", and perceived fatigue with the "Modified Borg Scale". Evaluations will be made before starting the exercise and at the end of the 8th week. Individuals in this group will participate in exercise sessions consisting of cognitive tasks combined with conventional exercises, 3 days a week, for a total of 8 weeks, under the supervision of a physical therapist. Each session will last approximately 40-50 minutes.
  Interventions: Device: Conventional exercises with dual task training (cognitive task)
- Action Observation Therapy (AOT) Group (Experimental): Cognitive functions will be assessed with the "Mini Mental State Test" and "Clock Drawing Test", balance and walking with the "Tinetti Balance and Walking Test", functional mobility with the "Timed Up and Go Test", muscle strength with a handheld dynanometer and "5-times chair sit-to-stand test", flexibility with the "sit-and-reach flexibility test", quality of life with the "CASP-19 Scale", and perceived fatigue with the "Modified Borg Scale". Evaluations will be made before starting the exercise and at the end of the 8th week. Individuals in this group will watch exercises on a computer screen in three sessions (in bed, sitting, and standing), three days a week for a total of eight weeks. Each exercise in each session will be monitored for two minutes, and each session will be performed under the supervision of a physical therapist for one minute. A one-minute break will be provided between sessions. Each session will last approximately 40-50 minutes.
  Interventions: Device: Conventional Exercise With Action Observation Therapy
- Control Group (CG) (Active Comparator): Cognitive functions will be assessed with the "Mini Mental State Test" and "Clock Drawing Test", balance and walking with the "Tinetti Balance and Walking Test", functional mobility with the "Timed Up and Go Test", muscle strength with a handheld dynanometer and "5-times chair sit-to-stand test", flexibility with the "sit-and-reach flexibility test", quality of life with the "CASP-19 Scale", and perceived fatigue with the "Modified Borg Scale". Evaluations will be made before starting the exercise and at the end of the 8th week. Individuals in this group will perform conventional exercise sessions under the supervision of a physiotherapist, 3 days a week, for a total of 8 weeks. (No action observation or cognitive tasks.) Each session will last an average of 40-50 minutes.
  Interventions: Device: Conventional Exercise (Control Group)

INTERVENTIONS:
Device: Conventional exercises with dual task training (cognitive task) — Individuals in this group will undergo exercise sessions under the supervision of a physiotherapist, with cognitive tasks added to conventional exercises, 3 days a week for a total of 8 weeks.
  EXERCISES
  1. Sit-Reach in Bed (15 seconds each)
  2. Hip Flexor Stretch Exercise (15 seconds each)
  3. Cat-Camel Exercise
  4. Bridge Exercise
  5. Biceps Curl/Triceps Extension/Upper Limb Abduction While Sitting in a Chair
  6. Sit-to-Stand in a Chair
  7. One-Legged Stand
  8. Mini Squat 9. Tandem Walk Cognitive Tasks to be Used in the Dual-Task Training Group Weeks 1 and 2 Simple single-digit addition Generate random numbers between 1 and 100 Count the days of the week Count the months of the year Repeat two spoken words Count from 0 to 100, incrementing by 10 Generate words starting with the specified letter Count from 1 to 100 The remaining cognitive task examples are in the study description. The exercises and cognitive tasks will be conducted sequentially and simultaneous
  Arms: Dual Task Training (DTT) Group
Device: Conventional Exercise With Action Observation Therapy — Individuals in this group will watch exercises on a computer screen in three sessions (in bed, sitting, and standing), three days a week for a total of eight weeks. Each exercise in each session will be monitored for two minutes, and each session will be performed under the supervision of a physical therapist for one minute. A one-minute break will be provided between sessions. Each session will last approximately 40-50 minutes. EXERCISES 1. Sit-Reach in Bed (15 seconds each) 2. Hip Flexor Stretch Exercise (15 seconds each) 3. Cat-Camel Exercise 4. Bridge Exercise 5. Biceps Curl/Triceps Extension/Upper Limb Abduction While Sitting in a Chair 6. Sit-to-Stand in a Chair 7. One-Legged Stand 8. Mini Squat 9. Tandem Walk For Example: After watching the video of the exercise period in which you sit and stand on a chair on the computer, do the same exercise by imitating it. (1 set, 10 repetitions) Device: Handheld dynanometer, chair, stopwatch, computer
  Arms: Action Observation Therapy (AOT) Group
Device: Conventional Exercise (Control Group) — Individuals in this group will perform conventional exercise sessions under the supervision of a physical therapist three days a week for a total of eight weeks. Each session will last approximately 40-50 minutes. No cognitive tasks or action monitoring therapy will be used during the exercises. EXERCISES 1. Sit-Reach in Bed (15 seconds each) 2. Hip Flexor Stretch Exercise (15 seconds each) 3. Cat-Camel Exercise 4. Bridge Exercise 5. Biceps Curl/Triceps Extension/Upper Limb Abduction While Sitting in a Chair 6. Sit-to-Stand in a Chair 7. One-Legged Stand 8. Mini Squat 9. Tandem Walk.
  Device: Handheld dynanometer, chair, stopwatch
  Arms: Control Group (CG)

SUMMARY:
Summary Aging leads to significant declines in both motor skills and cognitive functions. Declines in walking, balance, and general mobility are particularly evident, while declines in cognitive functions such as attention, memory, and decision-making are also observed. It is crucial to recommend therapeutic interventions that support healthy aging, aim to increase physical and cognitive function, and prevent physical limitations in individuals over 65. The aim of this study is to examine the effects of dual-task training and action observation therapy on parameters such as cognitive function, balance, gait, functional mobility, flexibility, strength, and quality of life in geriatric individuals. Sixty-six individuals over the age of 65 will be randomized into the Dual-Task Training (DTT) group (n=22), the Action Observation Therapy (EGT) group (n=22), and the Control Group (CG) (n=22), which will receive conventional exercise. The exercise program will be applied 3 days per week for 8 weeks in all three groups. To assess balance and walking, the "Tinetti Balance and Walk Test" will be used; to assess functional mobility, the "Timed Up and Go Test" will be used; to obtain information about muscle strength, the "Hand Dynanometer" and the "5-Time Chair Sit-to-Stand Test" will be used; the "Sit-and-Reach Flexibility Test" will be used; to assess quality of life, the "CASP-19 Quality of Life Scale for Elderly People - Turkey Version (CASP-13)" will be used; to assess cognitive functions, the "Mini Mental State Test" and the "Clock Drawing Test" will be used; and perceived fatigue levels after exercise will be assessed using the Modified Borg Scale. The analyses of the data taken into the study will be carried out using SPSS (Statistical Program in Social Sciences). The values of the data will be expressed as numbers, percentages, mean and standard deviation; the significance level (p) will be taken as 0.05 for comparison tests.

DETAILED DESCRIPTION:
Aging leads to significant declines in both motor skills and cognitive functions. While walking, balance, and general mobility are particularly impaired, cognitive functions such as attention, memory, and decision-making are also observed. The physical decline and cognitive decline associated with aging make it difficult for older adults to maintain independence in their daily activities. Studies have shown that cognitive impairments are directly related to mobility loss.

For individuals over 65, it is crucial to recommend therapeutic interventions that support healthy aging, aim to increase physical and cognitive function, and prevent physical limitations. In recent years, Action Observation Therapy (EGT), a cognitive strategy, has begun to be used in rehabilitation programs for the elderly, aiming to enhance motor learning and functional recovery. Action observation is a cognitive process based on observing actions performed by others without actually performing any movements. In EGT, participants first observe a meaningful action and then imitate it themselves. This stimulates motor learning and motor memory formation, facilitating the understanding and imitation of movements. EGT is a complementary strategy used to improve motor skills, facilitate motor learning, and stimulate neuroplasticity.

Another method used in recent years to improve motor skills and cognitive functions in the elderly is dual-task training (DTT). Dual-task training is based on the simultaneous execution of two motor-motor or cognitive-motor tasks. This methodology can be defined as the ability to simultaneously complete a secondary, cognitive, or motor task while maintaining the primary task of walking or postural balance.

A review of the literature has demonstrated that motor + cognitive dual-task training provided to elderly individuals is an effective intervention for improving cognitive function, health status, and life satisfaction, and reducing depression, in community-dwelling elderly individuals. Another study suggests that a dual-task intervention incorporating cognitive and physical activities in the elderly results in greater improvements in walking speed than interventions involving only physical activities. One study in the literature has reported that EGT improves cognitive function in individuals with MS. However, it appears that further research is needed on its effects on cognitive functions. A study published in 2025 reported that EGT, administered in addition to conventional treatment in elderly individuals, was effective in improving motor skills.

In light of this information, the investigators see that dual-task training and action observation therapy can be used to improve cognitive and physical functions in the elderly. However, it is also noteworthy that studies indicating that dual-task training can cause dual-task confusion in the elderly, leading to poorer performance. A review of the available literature reveals that studies on HDI and EGT mostly focus on a single disease, and no studies comparing these two methods, which may be effective in improving cognitive and motor functions in geriatric individuals, have been found.

More evidence is needed on outcome measures such as motor skills and cognitive functions for HDI and EGT in the geriatric population. Our proposed study will provide data and contributions to fill this gap in the literature.

Research question: In terms of the method used when implementing exercise programs in geriatric individuals, is conventional exercise training, dual-task training, or action observation therapy more effective on parameters such as cognitive functions, balance, walking, functional mobility, flexibility, strength, perceived effort, and quality of life?

Hypotheses:

H0a: Dual-task training applied to geriatric individuals does not improve cognitive functions, balance, walking, functional mobility, flexibility, strength, perceived effort, or quality of life.

H0b: Action observation therapy applied to geriatric individuals does not improve cognitive functions, balance, walking, functional mobility, flexibility, strength, perceived effort, or quality of life.

Hypothesis H0c: There is no difference between the groups in terms of the effects of conventional exercise training, dual-task training, and action observation therapy applied to geriatric individuals on cognitive functions, balance, walking, functional mobility, flexibility, strength, perceived effort, or quality of life.

Hypothesis H1a: Dual-task training applied to geriatric individuals improves cognitive functions, balance, walking, functional mobility, flexibility, strength, perceived effort, and quality of life.

Hypothesis H1b: Action observation therapy applied to geriatric individuals improves cognitive functions, balance, walking, functional mobility, flexibility, strength, perceived effort, and quality of life.

Hypothesis H1c: There is a difference between the groups in terms of the effects of conventional exercise training, dual-task training, and action observation therapy applied to geriatric individuals on cognitive functions, balance, walking, functional mobility, flexibility, strength, perceived effort, and quality of life.

Objectives: The aim of this study was to examine the effects of dual-task training and action observation therapy on parameters such as cognitive functions, balance, walking, functional mobility, flexibility, strength, perceived effort, and quality of life in geriatric individuals and to compare them with conventional exercise training.

Originality: There are studies demonstrating the use of dual-task training and action observation therapy to improve motor skills and cognitive functions in various diagnostic groups and in geriatric individuals. However, the investigators observe that there are more limited studies on the use of EGT in the elderly compared to HDI. The investigators believe that our study, which examines the effects of HDI and EGT on parameters such as motor skills and cognitive functions in geriatric individuals and compares these effects with conventional exercise training, will have a significant place in the literature. Our study aims to contribute to the literature by comparatively examining two different approaches that simultaneously intervene not only in motor skills but also in cognitive functions. Thus, it will provide insights into the holistic effects of different therapy methods on both motor skills and cognitive functions. The findings will provide recommendations for use in geriatric rehabilitation processes and help identify strategies that can improve overall health.

Type of Study This study is designed as a prospective experimental study. Location and Time of Study Data will be collected from nursing homes, nursing home elder care and rehabilitation centers, and Bahadın Elderly Living Center affiliated with the Ministry of Family and Social Services located in Yozgat and Çorum provinces. To avoid cross-contamination between the experimental and control groups, data for the experimental and control groups will be collected from different centers.

Research Population and Sample The sample for this study was determined using power analysis. According to calculations using the G*power 3.1.9.7 package program, with a total of 66 participants (22 in each group), an effect size of 0.40 and a significance level of 0.05, the power of the study will be 81.8%. This power is over 80%, making it sufficient. The sample will be selected from nursing homes, nursing home elder care and rehabilitation centers, and Bahadın Elderly Living Center affiliated with the Ministry of Family and Social Services located in Yozgat and Çorum provinces. These institutions will be listed, and three institutions will be selected from among the listed institutions, taking into account the high number of elderly individuals and their ability to meet the inclusion criteria. The groups to which geriatric individuals at these institutions will be assigned (HDE, EGT, and CG) will be determined using a sealed envelope method and randomized. Geriatric individuals at these institutions who meet the inclusion criteria and sign the informed consent form will be included in the study. A total of 66 participants will be selected, 22 geriatric individuals for each group.

Inclusion Criteria

* Agreeing to participate in the study
* Being over 65 years of age
* Scoring 24 or higher out of 30 on the Mini Mental State Examination
* Being literate Exclusion Criteria
* Having a musculoskeletal condition that prevents the performance of the tests and exercises
* Having a visual or hearing impairment that prevents participation in the study
* Having a neurological, psychiatric, or other condition that prevents participation in the study Having a medical diagnosis
* Having undergone any surgical procedure within the last six months Exclusion criteria
* The individual voluntarily withdraws from the study
* Failure to maintain exercise continuity (Participants must complete at least 80% of the exercise sessions (20/24 sessions) for the study to be considered applicable)
* Having an additional diagnosis that would prevent participation in exercise during the study period
* Failure to comply with instructions Data collection tools
* Sociodemographic Questionnaire
* Mini Mental State Examination (MMSE)
* Clock Drawing Test
* Tinetti Balance and Walking Test
* Timed Up and Go Test (TUG)
* Hand Dynamometer Grip Strength
* 5-Times Sit-to-Stand Chair Test (5KSOKT)
* Sit-and-Reach Flexibility Test
* CASP-19 Quality of Life Scale for Elderly People - Turkish Version (CASP-13)
* Modified Borg Scale (MBS) The sociodemographic characteristics of geriatric individuals will be determined with a descriptive questionnaire.

The outcome measures listed below will be assessed using the specified scales during the initial and final evaluations.

Assessment of Cognitive Functions: Because elderly individuals must have adequate communication and cognitive status, their cognitive functions will be assessed using the "Mini Mental State Examination (MMSE)" for inclusion in the study. The highest possible total score is 30, and scores below 24 indicate cognitive impairment. Volunteers scoring 24 or higher on the MMSE will be accepted into the study. The adapted Turkish version of this scale, originally known as the "Mini-Mental State Examination (MMSE), will be used. The MMSE will be used not only as an admission requirement but also in the final assessment. In addition, the "Clock Drawing Test" will be used to test constructional praxis, comprehension, and planning abilities. The individual is asked to draw a clock, place numbers inside it, and mark the time as it is announced. A score below four is consistent with impaired cognitive function. Scoring is as follows: Writing 12 in the correct place: 3 points, Writing all twelve numbers: 1 point, Drawing the hour and minute hands: 1 point, Marking the announced time correctly: 1 point.

Balance and Gait Assessment: The "Tinetti Balance and Gait Test (TDYT)" will be used to assess the balance and gait of geriatric individuals. The TDYT was first developed by Mary Tinetti under the name Performance-Oriented Assessment of Mobility Problems in Elderly Patients (POMA) to evaluate patients at high risk of falling. It was later developed and named the "Tinetti Gait and Balance Assessment". The TDYT evaluates balance ability and gait under two main headings. The first 9 questions are about balance, and the total score is the balance score. The next 7 questions are about gait, and the total score is the gait score. Three values are assigned for each unit: 0-1-2. 2 points represent correct performance of the specified movement; 1 point represents correct performance of the specified movement; A score of 0 indicates that the specified movement is performed with adaptations, and a score of 0 indicates that the movement cannot be performed. The sum of the balance and walking scores provides the total score. The total balance score is 16; a score below 11 indicates a risk of falling. The total walking score is 12; a score below 8 indicates a risk of falling. The Turkish validity and reliability study of the scale was conducted by Ağırcan.

Functional Mobility Assessment: The Timed Up and Go test (TUG) is a practical, equipment-free method that can be used to measure functional mobility in older individuals.

The individual being assessed stands up from a sitting position of approximately 46 cm, walks 3 meters, returns, and sits down again. The test is repeated twice. The elapsed time is measured in seconds .

Muscle Strength Assessment: Grip strength will be measured with a handheld dynamometer to obtain information about the general muscle strength of geriatric individuals. The study plans to measure hand muscle strength using a "Hand Dynamometer." During the measurement, the participant will be seated upright, as recommended by the American Association of Hand Therapists (AETD), and arm support will not be allowed on the sitting surface . Measurements will be performed three times, 10 seconds apart, and the average value will be used in the study. The measured force will be recorded in kg. Additionally, the "5-Time Chair Sit-to-Stand Test" (5KSOKT) will be used to assess lower extremity strength. In this test, the patient sits with their arms crossed over their shoulders and their back against a chair. On the "Start" command, the patient stands up and sits down quickly from a standard chair five times. The elapsed time is measured with a stopwatch .

Flexibility Assessment: The sit-and-reach flexibility test will be used to assess flexibility. The subject is seated on a flat surface, the soles of their bare feet are placed flat on the test bench, and then the subject is asked to extend their trunk forward as far as they can, holding the arms and fingers tense and straight for one or two seconds at the end position. After two attempts, the best score is recorded .

Quality of Life Assessment: The quality of life of geriatric individuals will be assessed using the "CASP-19 Elderly Quality of Life Scale - Turkish Version (CASP-13)." The CASP-19 Scale was developed by Hyde and colleagues to measure the quality of life of older adults. The CASP-13 Scale is the Turkish translation of the CASP-19 Scale and its adaptation for Turkish elderly. The validity and reliability study of the scale for Turkish elderly was conducted by Türkoğlu et al. The CASP-13 scale, the Turkish version of CASP-19, consists of 13 items. The questions are scored as 0 for "never," 1 for "occasionally," 2 for "sometimes," and 3 for "always." The scale score ranges from 0 to 39. A higher total score indicates an increase in quality of life. The positively worded items 3, 5, 6, 7, 8, 9, 10, 11, 12, and 13 constitute factor 1 (perception of autonomy and satisfaction), while the negatively worded and reverse-coded items 1, 2, and 4 constitute factor 2 (perception of disability). Cronbach's alpha coefficient of the scale was reported as 0.91. Assessment of Perceived Fatigue: Geriatric individuals' perceived fatigue levels after exercise will be assessed using the Modified Borg Scale (MBS). This scale was developed by Borg in 1970 to measure the effort expended during physical exercise . The MBS consists of 10 points indicating dyspnea severity. A score of 0 indicates no dyspnea or fatigue, while a score of 10 represents the highest degree of dyspnea and fatigue. Measurements will be taken after the first session of week 1 and the last session of week 8 for geriatric individuals in each group.

Study Design After obtaining informed consent for participation in the study, all participants, regardless of group, will undergo a pre- and post-intervention assessment by an experienced physiotherapist before group assignment. Following the pre-test assessments, patients will be informed about their groups and the relevant interventions will begin. The exercise program and cognitive tasks will be progressed every two weeks. The number of repetitions and sets will be adjusted as the exercise program progresses. Exercise sessions will be conducted three days per week for a total of eight weeks. Individuals in the HDI group will perform a cognitive task in addition to the conventional exercises. The cognitive tasks were determined based on a literature review. Individuals in this group will watch videos of exercises on a computer screen in three periods (in bed, sitting, and standing). Each exercise in each period will be viewed for 2 minutes and performed for 1 minute under the supervision of a physiotherapist. The EGT protocol was developed based on a review of literature. The CG will perform conventional exercises. Participants Geriatric individuals who meet the specified inclusion and exclusion criteria will be included in the study. Participants will be included in the study after signing a voluntary informed consent form.

Interventions Dual Task Training (DTT) Group: Individuals in this group will perform exercise sessions consisting of cognitive tasks combined with conventional exercises, 3 days a week, for a total of 8 weeks, under the supervision of a physiotherapist. Each session will last an average of 40-50 minutes.

Action Observation Therapy (EGT) Group: Individuals in this group will watch exercises on a computer screen in 3 periods (in bed, sitting, and standing). Each exercise in each period will be observed for 2 minutes and performed for 1 minute under the supervision of a physiotherapist. There will be a 1-minute break between periods. Each session will last an average of 40-50 minutes. Control Group (CG): Individuals in this group will perform conventional exercise sessions under the supervision of a physiotherapist three days a week for a total of eight weeks. Each session will last an average of 40-50 minutes.

Randomization In this study, to prevent any cross-contamination between the experimental and control groups, data for the experimental and control groups will be collected from different centers. To this end, after obtaining the necessary permits from the Ministry of Family and Social Services in Yozgat and Çorum provinces, and from the Bahadın Elderly Living Center in Yozgat province, the nursing homes, elderly care and rehabilitation centers, and elderly living centers in these provinces will be listed. Three institutions will be selected from the listed institutions, taking into account the large number of elderly individuals and whether they meet the inclusion criteria. The groups to which geriatric individuals in these institutions will be assigned-HDE, EGT, and CG-will be determined using a sealed-envelope method and randomized. Geriatric individuals who meet the inclusion criteria and sign the informed consent form will be included in the study. A total of 66 participants will be selected, 22 for each group, of whom 22 will be geriatric.

Exercise Protocol Based on the World Health Organization (WHO) exercise recommendations for older adults, the researcher has developed an exercise protocol suitable for participants over the age of 65, including balance, strengthening, and flexibility exercises performed in various positions, such as lying down, sitting, and standing. The exercises, prepared in accordance with World Health Organization recommendations, were developed by a physiotherapist experienced in geriatric rehabilitation. The exercise training program is designed to be performed three days a week. To facilitate patient comfort, the program will begin with exercises in the supine and prone positions and progress to exercises in the sitting and vertical positions. Each exercise session will consist of a warm-up (5 minutes); balance, flexibility, general muscle strengthening, and walking (30-40 minutes); and a cool-down (5 minutes). Each session will last 40-50 minutes.

Week 1: After randomization, the sample groups will be introduced. Information about the study will be provided. A seminar will be held on the benefits of physical activity in the elderly, and motivating individual training schedules will be presented to participants.

Week 2: Initial assessments of outcome measures will be conducted. Weeks 3-4: All three groups will begin training with warm-up exercises (5 minutes). Then, exercises including flexibility, strengthening, balance, and walking will begin (30-40 minutes). The session will conclude with cool-down exercises (5 minutes).

* DDT Group: They will complete the assigned exercises with cognitive tasks. For example: Counting the days of the week while doing sit-to-stand exercises in a chair (1 set, 10 repetitions).
* EGT Group: They will watch videos of the exercises in three periods before performing the assigned exercises. Each exercise in each period will be watched for 2 minutes, followed by 1 minute of that exercise. After a 1-minute break between each period, they will move on to the videos of the next period. For example: After watching a video of the period of the chair sit-and-stand exercise on the computer, perform the same exercise while imitating it. (1 set, 10 repetitions)
* CG: They will perform the specified exercises without any intervention. For example: Performing the chair sit-and-stand exercise (1 set, 10 repetitions) Weeks 5-6: All three groups will begin training with warm-up exercises (5 minutes). Then, they will begin exercises that include flexibility, strengthening, balance, and walking exercises (30-40 minutes). The session will conclude with cool-down exercises (5 minutes). The number of repetitions/sets will be progressive.
* DDT Group: They will complete the exercise with cognitive tasks while performing the specified exercises. For example: Counting the days of the week while performing the chair sit-and-stand (1 set, 12 repetitions)
* EGT Group: They will watch the exercise videos in three periods before performing the specified exercises. Each exercise in each period will be shown for 2 minutes, followed by 1 minute of that exercise. After a 1-minute break between each period, the participants will move on to the videos of the next period. For example: After watching the video of the period containing the chair sit-and-stand exercise on the computer, perform the same exercise while imitating it. (1 set, 12 reps)
* KG: They will perform the assigned exercises without any intervention. For example: Performing the chair sit-and-stand exercise (1 set, 12 reps) Weeks 7-8: All three groups will begin training with warm-up exercises (5 minutes). Then, they will begin exercises that include flexibility, strengthening, balance, and walking exercises (30-40 minutes). The session will conclude with cool-down exercises (5 minutes). The number of repetitions/sets will be progressive.
* DDT Group: They will complete the exercise with cognitive tasks while performing the assigned exercises. For example: Counting the days of the week while doing a chair sit-and-stand (2 sets, 10 repetitions).
* EGT Group: Before performing the designated exercises, they will watch videos of the exercises in three periods. Each exercise in each period will be watched for 2 minutes, followed by a 1-minute performance of that exercise. After a 1-minute break between each period, they will move on to the videos of the next period. For example: After watching the video of the period of the chair sit-and-stand exercise on the computer, they will perform the same exercise while imitating it. (2 sets, 10 repetitions).
* KG: They will perform the designated exercises without any intervention. For example: Performing the chair sit-and-stand exercise (2 sets, 10 repetitions).

Weeks 9-10: All 3 Groups will begin training with warm-up exercises (5 minutes). Then, they will begin performing exercises that include flexibility, strengthening, balance, and walking exercises (30-40 minutes). The session will conclude with a 5-minute cool-down exercise. The number of repetitions/sets will be progressive.

* DDT Group: They will complete the exercise with cognitive tasks while performing the assigned exercises. For example: Counting the days of the week while doing the chair sit-and-stand exercise (2 sets, 12 repetitions).
* EGT Group: They will watch videos of the exercises in three periods before performing the assigned exercises. Each exercise in each period will be watched for 2 minutes, followed by a 1-minute performance of that exercise, with a 1-minute break between each period before moving on to the videos of the next period. For example: After watching the video of the chair sit-and-stand exercise on the computer, they will perform the same exercise while imitating it. (2 sets, 12 repetitions).
* CG: They will perform the assigned exercises without any intervention. For example: Performing the chair sit-and-stand exercise (2 sets, 12 repetitions).

Week 11: Final assessments of outcome measures will be made. Pre-Exercise Warm-Up and Post-Exercise Cool-Down Exercises

Warm-Up Exercises (5 min)

* Side Stepping
* Touching the right and left legs while standing
* Reaching the arms to the right and left while standing
* Shoulder Rolls and Neck Movements Cool-Down Exercises (5 min)
* Step-Up
* Rotating the waist to the right and left with hands on hips
* Tightening and then relaxing the entire body while standing with eyes closed
* Shoulder Rolls and Neck Movements 8-Week Conventional Exercise Protocol to be Used in the Study EXERCISES

  1. Sit-Reach in Bed (15 seconds each)
  2. Hip Flexor Stretch Exercise (15 seconds each)
  3. Cat-Camel Exercise
  4. Bridge Exercise
  5. Biceps Curl/Triceps Extension/Upper Limb Abduction While Sitting in a Chair
  6. Sit-to-Stand in a Chair
  7. One-Legged Stand
  8. Mini Squat
  9. Tandem Walk Cognitive Tasks to be Used in the Dual-Task Training Group Weeks 1 and 2 Simple single-digit addition Generate random numbers between 1 and 100 Count the days of the week Count the months of the year Repeat two spoken words Count from 0 to 100, incrementing by 10 Generate words starting with the specified letter Count from 1 to 100 Say the digits of a 3-digit number in order Weeks 3 and 4 Simple double-digit addition Generate random odd and even numbers Count the days of the week in reverse Count the months of the year in reverse Repeat the three spoken words Count from 0 to 100 by increments of 5 Generate words starting with the specified letter and related to the specified category Say the even numbers between 1 and 100 in order Say the digits of a 4-digit number in order Weeks 5 and 6 Double-Digit Subtraction Generate random odd and even numbers between 1 and 100 Count the days of the week that start with a letter (e.g., the letter p) Count the months of the year that start with a letter (e.g., the letter e) Say three words, but ask them to repeat only the live ones Count backwards from 100 by 10s Generate words containing the two specified letters Say the odd numbers between 1 and 100 in order Say the digits of a 3-digit number in reverse order Weeks 7 and 8 Mixed addition and subtraction Add 1 to a random number, then say whether it is odd or even. When a day of the week is mentioned, say the previous and next day in order. When a month of the year is mentioned, say the previous and next month in order.

Say 3 words, but only repeat the vegetable words. Count backward from 100 by 5s. Generate words related to the specified category that contain 2 specified letters.

Say numbers between 1 and 100 whose sum is 10. Say the digits of a 4-digit number in reverse order.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the study
* Being over 65 years of age
* Scoring 24 or higher out of 30 on the Mini Mental State Examination
* Being literate

Exclusion Criteria:

* Having a musculoskeletal condition that would prevent the person from performing the tests and exercises.
* Having a vision or hearing impairment that would prevent participation in the study.
* Having a diagnosis of a neurological, psychiatric, or other condition that would prevent participation in the study.
* Having undergone any surgical procedure within the last six months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Tinetti Balance and Walking Test Score | From enrollment to the end of treatment at 8 weeks
  Participants' balance and walking performance will be assessed using the Tinetti Balance and Walking Test. The sum of the balance and walking scores provides the total score. The total balance score is 16; a score below 11 indicates a risk of falling. The total walking score is 12; a score below 8 indicates a risk of falling. Measurements will be taken before and at the end of the 8th week of Action Observation Therapy (AOT), Dual Task Training (DTT), and Control Group interventions, and comparisons will be made between the groups.
Timed Up and Go Test Score | From enrollment to the end of treatment at 8 weeks
  Functional mobility will be measured in seconds with the Timed Up and Go (TUG) test. The participant rises from a chair, walks 3 meters, turns, and sits back down. Elapsed time is measured in seconds. Measurements will be taken before and after the Action Observation Therapy (AOT), Dual Task Training (DTT) and Control Group interventions, and at the end of the 8th week, for comparison between groups.
Mini Mental State Examination (MMSE) Test Scores | From enrollment to the end of treatment at 8 weeks
  Participants' general cognitive status will be evaluated with the Mini Mental State Examination (MMSE) Test. The highest possible total score on the mini mental test is 30, and scores below 24 indicate cognitive impairment. Measurements will be taken before and 8 weeks after the Action Observation Therapy (AOT), Dual Task Training (DTT), and Control Groups, and will be compared.
Clock Drawing Test Score | From enrollment to the end of treatment at 8 weeks
  Participants' executive functions, visual-spatial skills and planning ability will be evaluated with the Clock Drawing Test. In the clock drawing test, a score below four is consistent with impaired cognitive function. Measurements will be taken before and 8 weeks after the Action Observation Therapy (AOT), Dual Task Training (DTT), and Control Groups, and will be compared.
Hand dynamometer Score | From enrollment to the end of treatment at 8 weeks
  Grip strength will be measured with a hand dynamometer. Measurements will be taken before and after 8 weeks of action observation therapy (AOT), dual-task training (DDT), and the Control Group for comparison. The measurement will be taken three times, 10 seconds apart, and the average value will be used in the study. The measured force will be recorded in kg.
5-times chair sit-to-stand test score | From enrollment to the end of treatment at 8 weeks
  To measure lower extremity muscle strength, the participant will be asked to sit down and stand up from a chair five times in a row using a sit-to-stand test. The time will be recorded in seconds. Measurements will be taken before and after 8 weeks of action observation therapy (AOT), dual-task training (DDT), and the Control Group for comparison.
Sit-Reach Test Score | From enrollment to the end of treatment at 8 weeks
  Flexibility will be assessed with the sit-and-reach test. The participant's forward reach while sitting will be measured in cm. Measurements will be taken before and after eight weeks of action observation therapy (AOT), dual-task training (DDT), and the control group, and for intergroup comparisons.
CASP-19 Elderly Quality of Life Scale-Turkish Version (CASP-13) Score | From enrollment to the end of treatment at 8 weeks
  Participants' quality of life will be assessed using the CASP-19 Elderly Quality of Life Scale-Turkish Version (CASP-13). Scale scores range from 0 to 39. Higher total scores indicate improved quality of life. Measurements will be taken before and 8 weeks after interventions in the action observation therapy, dual-task training, and control groups. Measurement results will be compared across groups.
Modified Borg Scale (MBS) Score | From enrollment to the end of treatment at 8 weeks
  Geriatric individuals' perceived fatigue levels after exercise will be assessed using the Modified Borg Scale (MBS). The MBS consists of 10 points indicating dyspnea severity. A score of 0 indicates no dyspnea or fatigue, while a score of 10 indicates the highest degree of dyspnea and fatigue. Measurements will be taken after the first session of week 1 and the last session of week 8 for geriatric individuals in the action observation therapy, dual-task training, and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Gül Turan, Lecturer, Principal Investigator — Inonu University; Fatma Kızılay, Associate Professor, Study Director — Inonu University
Locations (1):
- In the provinces of Yozgat and Çorum, 3 institutions will be selected among the nursing homes, nursing homes and rehabilitation centers affiliated with the Ministry of Family and Social Services + Bahadın Elderly Living Center., Yozgat, Yozgat / Central, Turkey (Türkiye)

REFERENCES:
- [Background] Syrigos KN, Karayiannakis AJ, Zbar A. Mucins as immunogenic targets in cancer. Anticancer Res. 1999 Nov-Dec;19(6B):5239-44. PMID 10697542
- [Background] Smeyers-Verbeke J, Verbeelen D. Determination of aluminum in bone by atomic absorption spectroscopy. Clin Chem. 1985 Jul;31(7):1172-4. PMID 4006186
- [Background] McKibbin EC, Wilson KG. Affairs of the heart: patients' personal constructions of a cardiac event and their effect on lifestyle change. Curationis. 2001 Mar;24(1):31-9. doi: 10.4102/curationis.v24i1.796. PMID 11885144
- [Background] Stuart RK, McDonald JW, Ahuja SP, Coles JC. Platelet survival in patients with prosthetic heart valves. Am J Cardiol. 1974 Jun;33(7):840-4. doi: 10.1016/0002-9149(74)90630-4. No abstract available. PMID 4597816
- [Background] Del Fante P, Jenniskens F, Lush L, Morona D, Moeller B, Lanata CF, Hayes R. HIV, breast-feeding and under-5 mortality: modelling the impact of policy decisions for or against breast-feeding. J Trop Med Hyg. 1993 Aug;96(4):203-11. PMID 8345538
- [Background] Kimura M, Tohya K, Toda S. An electron microscopical observation of the endoneurial mast cells of the laboratory musk shrew: Suncus murinus). Anat Anz. 1988;165(2-3):143-50. PMID 3400880
- [Background] Demirtas Karaoba D, Talu B. The Effect of Video-Based Action Observation Training and Live Action Observation Training on Motor Function, Activity Participation, and Secondary Outcome Measures in Children With Spastic Diparetic Cerebral Palsy: A Randomized Controlled Study. J Child Neurol. 2024 Nov;39(13-14):470-480. doi: 10.1177/08830738241280838. Epub 2024 Oct 8. PMID 39376091
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Hyde M, Wiggins RD, Higgs P, Blane DB. A measure of quality of life in early old age: the theory, development and properties of a needs satisfaction model (CASP-19). Aging Ment Health. 2003 May;7(3):186-94. doi: 10.1080/1360786031000101157. PMID 12775399
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Tinetti ME. Performance-oriented assessment of mobility problems in elderly patients. J Am Geriatr Soc. 1986 Feb;34(2):119-26. doi: 10.1111/j.1532-5415.1986.tb05480.x. No abstract available. PMID 3944402
- [Background] Stahelin HB, Monsch AU, Spiegel R. Early diagnosis of dementia via a two-step screening and diagnostic procedure. Int Psychogeriatr. 1997;9 Suppl 1:123-30. doi: 10.1017/s1041610297004791. PMID 9447435
- [Background] Baek CY, Chang WN, Park BY, Lee KB, Kang KY, Choi MR. Effects of Dual-Task Gait Treadmill Training on Gait Ability, Dual-Task Interference, and Fall Efficacy in People With Stroke: A Randomized Controlled Trial. Phys Ther. 2021 Jun 1;101(6):pzab067. doi: 10.1093/ptj/pzab067. PMID 33611557
- [Background] Rocca MA, Meani A, Fumagalli S, Pagani E, Gatti R, Martinelli-Boneschi F, Esposito F, Preziosa P, Cordani C, Comi G, Filippi M. Functional and structural plasticity following action observation training in multiple sclerosis. Mult Scler. 2019 Oct;25(11):1472-1487. doi: 10.1177/1352458518792771. Epub 2018 Aug 7. PMID 30084706
- [Background] Leone C, Feys P, Moumdjian L, D'Amico E, Zappia M, Patti F. Cognitive-motor dual-task interference: A systematic review of neural correlates. Neurosci Biobehav Rev. 2017 Apr;75:348-360. doi: 10.1016/j.neubiorev.2017.01.010. Epub 2017 Jan 16. PMID 28104413
- [Background] Winser SJ, Chan HTF, Ho L, Chung LS, Ching LT, Felix TKL, Kannan P. Dosage for cost-effective exercise-based falls prevention programs for older people: A systematic review of economic evaluations. Ann Phys Rehabil Med. 2020 Jan;63(1):69-80. doi: 10.1016/j.rehab.2019.06.012. Epub 2019 Jul 12. PMID 31306811